CLINICAL TRIAL: NCT04380116
Title: Preliminary Effectiveness of Remotely Monitored Blood Alcohol Concentration Device as Treatment Modality
Acronym: Soberlink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Frank D Buono, PHD, Associate Research Scientist, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000027787
Record Dates: First submitted 2020-04-29; First posted 2020-05-08 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Sb+Aware (Experimental): Patients will access to the Soberlink device and receive treatment with Aware Recovery Care
  Interventions: Device: Soberlink
- Aware (No Intervention): Patients will only have access to Aware Recovery Care

INTERVENTIONS:
Device: Soberlink — Soberlink is a comprehensive alcohol monitoring system designed to remotely monitor a person's Blood Alcohol Concentration (BAC). Combining a professional grade handheld breathalyzer with wireless connectivity, the technology includes real-time facial recognition, robust tamper detection and real-time alerting.
  Arms: Sb+Aware

SUMMARY:
State the scientific aim(s) of the study, or the hypotheses to be tested. The purpose of the current study is to evaluate the usage and acceptability of the Soberlink's blood alcohol concentration (BAC) unit in collaboration with Aware treatment to assess increased sobriety within patients suffering from alcohol use disorder (AUD).

The specific AIMS will be:

1. To determine the effectiveness of Soberlink's ability to increase abstinence
2. To evaluate the impact of Soberlink's device on the participant based on their quality of health and sobriety.
3. To evaluate the extent to which need for higher levels of follow-up care and treatment is reduced for individuals who have had access to the Soberlink device.

ELIGIBILITY:
Inclusion Criteria:

* are at least 21 years old,
* currently enrolled at Aware In home treatment,
* Primary or secondary DSM-5 diagnosis of alcoholism use disorder (AUD).

Exclusion Criteria:

* Current suicide or homicide risk,
* meet criteria for DSM-IV current psychotic disorder, or bipolar disorder,
* does not have phone access with text message capabilities
* Unable to read or understand English,
* Unable to complete the study because of anticipated incarceration or move,
* Life-threatening or unstable medical problems,
* No course of current or pending legal action,
* Soberlink results being used for child custody or legal circumstance.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aware Recovery Care, North Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buono FD, Gleed C, Boldin M, Aviles A, Wheeler N. Preliminary Effectiveness of a Remotely Monitored Blood Alcohol Concentration Device as Treatment Modality: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Jan 14;11(1):e30186. doi: 10.2196/30186. PMID 35029534
- See also: Related Info — http://www.soberlink.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sb+Aware | Aware
Started | 48 | 48
Completed | 43 | 32
Not Completed | 5 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sb+Aware | Aware | Total
Number analyzed (Participants) | 43 | 32 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (10.5) | 44.1 (11.8) | 45.04 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 57
  Male | 13 | 5 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 22 | 56
  Black or African American | 3 | 4 | 7
  Hispanic | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 43 | 32 | 75
Marital Status [Count of Participants; unit: Participants]
  Single | 5 | 9 | 14
  Married | 26 | 19 | 45
  Divorced | 10 | 1 | 11
  Separated | 2 | 2 | 4
  Widowed | 0 | 1 | 1
Highest Level of Education Completed [Count of Participants; unit: Participants]
  High School | 11 | 9 | 20
  Some College | 5 | 6 | 11
  Associates | 1 | 1 | 2
  Bachelors | 12 | 10 | 22
  Advanced Degree | 14 | 6 | 20
Work Status [Count of Participants; unit: Participants]
  Employed | 33 | 27 | 60
  Student | 1 | 0 | 1
  Retired | 3 | 2 | 5
  Unemployed | 6 | 3 | 9
Generalized Anxiety Disorder-7 questionnaire [Mean (Standard Deviation); unit: score on a scale] — Generalized Anxiety Disorder-7 questionnaire is a 7-item validated questionnaire used to screen for anxiety with a range of scores from 0-3. A cumulative score of ≥8 is considered positive for anxiety with lower scores indicating no or mild anxiety. Minimum score is 0 and the maximum score 21. Total score was provided.
  score on a scale | 14.8 (4.3) | 15.3 (6.1) | 15.1 (5.8)
Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — PHQ-9 is a 9-item validated questionnaire used to screen for depression with a range of scores from 0-45. A cumulative score of ≥10 is considered positive with lower scores indicating no or mild anxiety.
  units on a scale | 13.3 (5.5) | 12.6 (4.8) | 12.9 (5.8)
Previous Alcohol Treatments [Mean (Standard Deviation); unit: mean number of participants] — Mean number of participants that have had previous treatment for Alcohol. Data was extracted from self-reported demographic information by the participant.
  mean number of participants | 3.1 (2.2) | 2.9 (1.8) | 3.02 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Time Line Follow Back (TLFB)
Description: The Alcohol TLFB is a drinking assessment method that obtains estimates of daily drinking and has been evaluated with clinical and nonclinical populations.
  Using a calendar, people provide retrospective estimates of their daily drinking over a specified time (previous month). The Alcohol TLFB allows several dimensions of a person's drinking to be separately examined: (a) variability (i.e., scatter); (b) pattern (i.e., shape); and (c) extent of drinking (i.e., elevation; how much).
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: drinks per month
Arm/Group | Sb+Aware | Aware
Number analyzed (Participants) | 43 | 32
drinks per month | 27.1 (2.2) | 21 (3.1)

2. Secondary Outcome: Quality of Life Survey
Description: the quality of life survey (QLS) is a 16 question self-directed 7-point likert based survey (7-delighted; 1-terrible. The total score is 112, and the lowest is 16. Generally higher score indicate better QLS.
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sb+Aware | Aware
Number analyzed (Participants) | 43 | 32
score on a scale | 73.53 (26.3) | 75.9 (23.2)
Statistical Analysis 1: Comparison: Sb+Aware vs Aware; Test type: Superiority; p = .366, ANOVA

3. Secondary Outcome: Mean Positive BAC Response With Soberlink
Description: sensor to detect alcohol levels at an accuracy of +/-.005 BAC. BAC is established by the manufacturer based on predetermined cut off points. Mean number of positive responses, recorded using Soberlink sensor.
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: Positive responses
Arm/Group | Sb+Aware
Number analyzed (Participants) | 43
Positive responses | 1.09 (1.4)

4. Secondary Outcome: Alcohol Abstinence Self-efficacy Scale for Temptation.
Description: Alcohol Abstinence Self-Efficacy Scale for Temptation is a 5 item 5 point Likert scale questionnaire where 0 indicates not at all, and 4 indicates extremely, total score has a range between 0-80. Lower scores indicate that participants do not believe they can resist the temptation to drink alcohol
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sb+Aware | Aware
Number analyzed (Participants) | 43 | 32
score on a scale | 20.5 (18.5) | 20.1 (19.4)

5. Secondary Outcome: Alcohol Abstinence Self-efficacy Scale for Confidence
Description: Alcohol Abstinence Self-Efficacy Scale for Confidence is a 5 item 5 point Likert scale questionnaire where 0 indicates not at all, and 4 indicates extremely, total score has a range between 0-80. Higher scores indicate higher confidence in abstaining from alcohol.
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sb+Aware | Aware
Number analyzed (Participants) | 43 | 32
score on a scale | 50.2 (27.5) | 46.3 (27.1)

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Arm/Group | Sb+Aware | Aware
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/32
Other Adverse Events (participants affected / at risk) | 0/43 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT04380116/Prot_SAP_000.pdf